CLINICAL TRIAL: NCT03173287
Title: Quantification of Hepatic Fibrosis by IVIM Sequences in 1.5T MRI.
Acronym: IVIM-MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-327; 2016-A02066-45 (Other: 2016-A02066-45)
Record Dates: First submitted 2017-05-09; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Liver Fibrosis; MRI; IVIM; Liver Biopsy
Keywords: Hepatic fibrosis; IVIM; 1.5T MRI
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hepatic biopsy (Experimental): The patients having benefited from a hepatic biopsy for evaluation of the hepatic fibrosis, will benefit in 10 days of a MRI in the service of radiology of the hospital Gabriel Montpied.
  Interventions: Procedure: Quantification of liver fibrosis

INTERVENTIONS:
Procedure: Quantification of liver fibrosis — Procedure MRI and liver biopsy

SUMMARY:
Quantification of hepatic fibrosis by IVIM sequences in 1.5T MRI.

DETAILED DESCRIPTION:
Early and accurate diagnosis of hepatic fibrosis in patients with chronic liver disease is essential and essential. This assessment could be performed by a non-invasive MRI method.

The main objective of this study is to show that the measured perfusion-related scattering value (D *) is related to the hepatic fibrosis stage.

Secondary objectives

* Evaluation of infusion fraction (f) and fibrosis stage.
* Evaluation of molecular diffusion (D) and fibrosis stage.
* Evaluation of ADC and fibrosis stage.
* Assess whether there is a link between the etiology of fibrosis and the value of the diffusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatic biopsy (trans-parietal or trans-jugular) in the context of liver disease
* Signature of written consent

Exclusion Criteria:

* Contra-indications to MRI
* Refusal of protocol
* Underage patients and protected adults

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Measured perfusion-related scattering value | at day 1
  The main objective of this study is to show that the measured perfusion-related scattering value (D *) is related to the hepatic fibrosis stage.

SECONDARY OUTCOMES:
Measured perfusion-related of infusion fraction | at day 1
Measured perfusion-related of molecular diffusion | at day 1
Measured perfusion-related of ADC | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Benoit MAGNIN, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France